CLINICAL TRIAL: NCT05351242
Title: Thermotherapy Against Persistent Bacterial LUNG Infections
Acronym: THERM-A-LUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THERM-A-LUNG
Record Dates: First submitted 2022-04-19; First posted 2022-04-28 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Lung Diseases, Obstructive; Bronchiectasis; Asthma; Copd; Chronic Obstructive Pulmonary Disease; Chronic Lung Infections
MeSH Terms: conditions — Lung Diseases, Obstructive; Bronchiectasis; Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermotherapy/sauna bath (Experimental): Must go to a sauna (min. Temperature 85℃) min. 4 times a week for 6 months. Each sauna bath must last at least 7 minutes. The intervention patients receive a subscription card for a sauna during the period. Patients will still receive pre-existing treatment
  Interventions: Other: Thermotherapy/sauna bath
- No thermotherapy/sauna bath (No Intervention): Not allowed to go to a sauna for 6 months. Patients who come to do so, by e.g. an oversight, however, remain in the study, to avoid introducing bias. It will be registered as a "protocol violation", but the patient will be included in Intention To Treat analysis and modified Intention To Treat analysis. Patients will still receive pre-existing treatment.

INTERVENTIONS:
Other: Thermotherapy/sauna bath — Thermotherapy/sauna bath
  Arms: Thermotherapy/sauna bath

SUMMARY:
The aim of this study is to determine whether an intervention with frequent thermotherapy will be able to reduce the amount of colonizing bacteria in the bronchoalveolar lavage sample and eradicate the colonizing bacteria.

DETAILED DESCRIPTION:
Normally, bacterial lung infections are acute such as community-acquired pneumonia and typically resolve after antibiotic therapy without leaving much lasting damage on the lungs. However, a great amount of persons with disrupted clearance of mucus and/or lung immune system get persistent lung infections, which can be life-long, usually do not resolve even with antibiotics, and can greatly increase morbidity and mortality. IThese persistent lung infections are thus characterized by stable periods with exacerbations inbetween, akin to chronic lung diseases such as asthma, chronic obstructive pulmonary disease (COPD) and bronchiectasis. In addition, it has not been thoroughly investigated whether antibiotic regimens have an effect on disease control, as biofilm formation prevents antibiotics from killing the bacteria.

This is a randomized, controlled, multi-center, superiority trial evaluating the effect of a thermotherapy intervention, consisting of min. 7 minutes stay in min. 85℃ environment at least 4 times a week for 6 months, in persons with persistent bacterial lung infection, defined as min. 2 positive cultures during the last 24 months for one of the following bacteria: Pseudomonas aeruginosa, Achromobacter xylosoxidans, Stenotrophomonas maltophilia, Klebsiella oxytoca, Klebsiella pneumoniae, Haemophilus influenzae or Staphylococcus aureus, incl. 1 positive culture after attempted eradication therapy. The aim of the study is to investigate whether thermotherapy may offer a valid proposal for treatment of chronic lung infections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Competent and capable
* FEV1>1,0 L
* Have had a positive culture from sputum or BAL min. 2 times in the last 24 months for bacteria of the species: Pseudomonas aeruginosa, Stenotrophomonas maltophilia, Staphylococcus aureus, Haemophilus influenzae, Achromobacter xylosoxidans, Klebsiella oxytoca or Klebsiella pneumoniae. In addition, min. 1 positive culture after treatment with antibiotics
* Willing to go to a sauna (min. temperature of 85℃ for at least 7 minutes) four times weekly for six months or avoid going to a sauna for six months

Exclusion Criteria:

* Allergy to lidocaine and/or midazolam
* Contraindications to bronchoscopy
* Previous severe laryngospasm (intubation requiring)
* Pregnancy/breastfeeding
* Severe linguistic problems or inability to give informed consent
* Severe mental illness that is not controlled with medication. NB: Patients with controlled mental illness can be included and will be asked on an equal footing as others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in bacterial growth (measured in cfu/mL) from bronchoalveolar lavage after 6 months | 6 months
Eradication of the cultured bacteria at baseline, defined by no use of antibiotics the last 14 days at the follow-up assessment after 6 months | 6 months

SECONDARY OUTCOMES:
Number of hospitalizations for all causes or death within 6 months | 6 months
Number of antibiotic treatment regimes within 6 months | 6 months
Physical performance measured by distance walked over 6 minutes | 6 months
Changes in FEV1 after 6 months | 6 months
Changes in BMI after 6 months | 6 months
Clinically relevant changes in Chronic Obstructive Pulmonary Disease Assessment Test-score (range from 0-40, higher is worse) after 6 months | 6 months
Changes in status from Medical Research Council-dyspnea score (range from 0-5, higher is worse) from <3 to 3≥, after 6 months | 6 months
Changes in composition of the lung microbiota after 6 months | 6 months
Changes in abundance of the lung microbiota after 6 months | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte University hospital, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP